CLINICAL TRIAL: NCT04798040
Title: Effects of Lavender Aromatherapy and Cold Application on Pain During Drain Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Cemile Celebi, Principle Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20012021-2/IV
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Major Abdominal Surgery
Keywords: lavender oil; aromatherapy; cold application; pain; nursing care; drain removal
MeSH Terms: conditions — Pain | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Routine treatment and nursing care of the clinic will be applied to the patients without any application.
  Routine interventions applied to the control group during silicone drain removal in the clinic:
  1. The patient will be informed about the procedure.
  2. The consent of the patient who agrees to participate in the study will be obtained.
  3. The patient will mark the pain he feels due to the silicone drain on the Numeric Rating Scale .
  4. The patient will mark the pain again from the Numeric Rating Scale immediately after the procedure.
  5. The patient will fill the Numeric Rating Scale 15 minutes after the removal of the silicone drain.
- Cold application group (Experimental): The patient will mark the pain he feels due to the silicone drain on the Numeric Rating Scale. A gel pad with a temperature of -10 ° C and a homogeneous distribution when cooled will be placed so that the patient is in full contact with the silicone drain.Since the skin temperature must fall below 13.6 ° C for cold application to have a local analgesic effect, the application will be terminated when the patient's skin temperature is 13.6 ° C by measuring every one minute during the cold application and the physician will be informed that the patient is ready.The patient will mark the pain again from the Numeric Rating Scale immediately after the procedure. The patient will fill the Numeric Rating Scale15 minutes after the removal of the silicone drain.
  Interventions: Other: cold application
- Lavender oil group (Experimental): All patients who accept the study will be tested for lavender oil before the procedure to exclude sensitivity to lavender. Patients in the lavender group will be given oxygen with a lavender oil covered face mask 15 minutes before the silicone drain is removed. Two drops of 2% lavender oil will be applied with a cotton swab inside the oxygen face mask.
  The patient will mark the pain he feels due to the silicone drain on the Numeric Rating Scale.The patient will mark the pain again from the Numeric Rating Scale immediately after the procedure.The patient will fill the Numeric Rating Scale 15 minutes after the removal of the silicone drain.
  Interventions: Other: lavender oil inhalation
- Oxygen administration (Experimental): The patient will be informed about the procedure. Consent of the patient who agrees to participate in the study will be obtained. Patients in the oxygen administration group will be given 2 lt/min oxygen with a face mask 15 minutes before the silicone drain is removed. The patient will mark the pain he feels due to the silicone drain on Numeric Rating Scale. The patient will re-mark the pain from Numeric Rating Scale immediately after the procedure. The patient will fill the Numeric Rating Scale 15 minutes after the removal of the silicone drain. Before the procedure, as soon as the procedure is over and 15 minutes after the procedure, the patient's vital signs will be measured.
  Interventions: Other: oxygen administration

INTERVENTIONS:
Other: cold application — To reduce pain, cold application is applied around the drain before the drain is removed.
  Arms: Cold application group
Other: lavender oil inhalation — To reduce pain, lavender oil is inhaled prior to drain removal.
  Arms: Lavender oil group
Other: oxygen administration — To reduce pain, oxygen is inhaled prior to drain removal.
  Arms: Oxygen administration

SUMMARY:
This study evaluates the effect of lavender aromatherapy and cold application on pain during drain removal. The investigators hypothesize that there is no difference in pain prevention between lavender oil inhalation and local cold application.

DETAILED DESCRIPTION:
It is common practice to place a drainage tube in the peritoneal cavity after abdominal surgery. Although drain application is an important initiative, the severe pain caused during the removal process should also be controlled . Pain and discomfort continue to be a problem during the removal of surgical silicone drains. In the literature, patients describe silicone drain removal as a very painful procedure. Analgesics applied during drain removal are among the commonly used methods in the treatment of acute pain . However, the fact that the response of the patient to pharmacological treatment is variable and the pain cannot be completely controlled with these agents necessitates the use of non-pharmacological methods in addition to pharmacological agents in the control of severe pain.

One of the non-pharmacological methods used in pain control is cold application. Cold application reduces the oxygen and nutrient requirement of tissues by slowing down metabolism, and eliminates pressure and tension on nerve endings by limiting inflammation, spasm and edema; It creates an analgesic effect by slowing or blocking the conduction velocity of peripheral nerves. In addition, it increases the release of endogenous opioids by stimulating the touch receptors with the gate-control mechanism, thereby reducing pain.

Aromatherapy using essential oils is now used by many healthcare professionals in the UK, Australia, Canada, New Zealand, Germany and Switzerland as a part of patient care to reduce pain and stress. When the effects of essential oils used for this purpose are examined; It is seen that it accelerates blood and lymph circulation, relieves muscle spasm and has calming effects. It is reported that these effects of essential oils are both absorbed from the skin and stimulated the sense of smell. In the literature, it is emphasized that some known or unknown analgesic components in oils affect the release of substances such as dopamine, endorphin, noradrenaline and serotonin in the brain stem, and that they have analgesic properties that are said to be formed as a result.

The physiological and psychological effects of aromatherapy have long been known in complementary medicine. Lavender oil has been associated with its mood enhancing and analgesic properties in healthy subjects and experimental nociception. This therapy has been successfully used in clinical settings to alleviate a wide variety of pain, such as dressing change in the intensive care unit, palliative care, for the control of labor pain, and chronic pain. There are numerous studies describing the use of this therapy to relieve anxiety and improve mood. Limited studies have shown that aromatherapy is beneficial for women who give birth and reduces the need for pain medication.

Considering the potential positive effect of lavender oil on the physiological and psychological state of the patient and the positive effect of cold application on the pain mechanism, our study was planned to determine the effectiveness of lavender aromatherapy and cold application in controlling the pain that occurs during the drain removal process.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-80,
* Being conscious, oriented and cooperative,
* Can speak and understand Turkish,
* After the surgery with silicone drains
* General condition stable,
* Patients who received written and verbal consent to participate in the study will be included.

Exclusion Criteria:

* Patients with asthma, bronchitis, chronic obstructive pulmonary disease
* Patients with contact dermatitis against cosmetic fragrances
* Patients who are pregnant
* Patients with poor general condition
* Oriented, non-cooperative patients
* Patients whose consent is not taken will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Pain level before the drain removal | 15 minutes before the drain removal
  Pain scores of all patients (lavender oil, cold application, oxygen administration and control group) before removal of the drain were evaluated using the Numerical Rating Scale (NRS). The Numeric Rating Scale is used to digitize the level of pain that cannot be measured numerically. In this scale, patients are asked to describe their pain by numbers, with "0" for painlessness and "10" for the highest unbearable pain. According to this scoring system, less than 3 points indicate mild pain, 3-6 points indicate moderate pain, and more than 6 points indicate severe pain.
Pain level as soon as the drain removal | as soon as the drain is removed.
  As soon as the drain was removed, the pain scores of all patients (lavender oil, cold application, oxygen administration and control group) were evaluated using the Numerical Rating Scale (NRS). The Numeric Rating Scale is used to digitize the level of pain that cannot be measured numerically. In this scale, patients are asked to describe their pain by numbers, with "0" for painlessness and "10" for the highest unbearable pain. According to this scoring system, less than 3 points indicate mild pain, 3-6 points indicate moderate pain, and more than 6 points indicate severe pain.
Pain level after drain removal | 15 minutes after the drain is removed
  After the drain was removed, the pain scores of all patients (lavender oil, cold application, oxygen administration and control group) evaluated using the Numerical Rating Scale (NRS). The Numeric Rating Scale is used to digitize the level of pain that cannot be measured numerically. In this scale, patients are asked to describe their pain by numbers, with "0" for painlessness and "10" for the highest unbearable pain. According to this scoring system, less than 3 points indicate mild pain, 3-6 points indicate moderate pain, and more than 6 points indicate severe pain.

SECONDARY OUTCOMES:
Oxygen Saturation (SPO2) before drain removal | 15 minutes before the drain removal
  Before the drain removal oxygen saturation level (SPO2) (percent) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. The researcher measured the oxygen saturation in subcutaneous arterial blood with a "Pulse oximeter" device that is reliable, easy to use, does not require calibration and does not cause pain to the patient in its application. Normal value of oxygen saturation (SpO2) (percent) was accepted as 96-98%. After placing a probe in the periphery (on the patient's finger) by the investigator, the signal received from the periphery and the value on the image screen (monitor) where the pulse wave sample was projected was recorded as oxygen saturation.
Oxygen Saturation (SPO2) as soon as the drain removal | as soon as the drain removal
  As soon as the drain removal, the oxygen saturation level (SPO2) (percent) of all patients (lavender oil, cold application, oxygen administration and control group) was measured.The researcher measured the oxygen saturation in subcutaneous arterial blood with a "Pulse oximeter" device that is reliable, easy to use, does not require calibration and does not cause pain to the patient in its application. Normal value of oxygen saturation (SpO2) (percent) was accepted as 96-98%. After placing a probe in the periphery (on the patient's finger) by the investigator, the signal received from the periphery and the value on the image screen (monitor) where the pulse wave sample was projected was recorded as oxygen saturation.
Oxygen Saturation (SPO2) after the drain removal | 15 minutes after the drain is removed
  After the drain removal oxygen saturation level (SPO2)(percent) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. The researcher measured the oxygen saturation in subcutaneous arterial blood with a "Pulse oximeter" device that is reliable, easy to use, does not require calibration and does not cause pain to the patient in its application. Normal value of oxygen saturation (SpO2) (percent) was accepted as 96-98%. After placing a probe in the periphery (on the patient's finger) by the investigator, the signal received from the periphery and the value on the image screen (monitor) where the pulse wave sample was projected was recorded as oxygen saturation.
Systolic and Diastolic Blood Pressure before the drain removal | 15 minutes before the drain removal
  Before the drain removal blood pressure (mm/Hg) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. Blood Pressure Measurement was performed using a conventional cuffed sphygmomanometer that can measure systolic and diastolic blood pressure, whose reliability was approved according to international standards and calibrated by the company in technical laboratories for certain periods. The cuff of the sphygmomanometer will be inflated to 20 mm / Hg above the systolic pressure by tying it to cover 2/3 of the arm, and the measurement will be carried out by the researcher.
Systolic and Diastolic Blood Pressure as soon as the drain removal | as soon as the drain removal
  As soon as the drain removal blood pressure (mm/Hg) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. Blood Pressure Measurement was performed using a conventional cuffed sphygmomanometer that can measure systolic and diastolic blood pressure, whose reliability was approved according to international standards and calibrated by the company in technical laboratories for certain periods. The cuff of the sphygmomanometer will be inflated to 20 mm / Hg above the systolic pressure by tying it to cover 2/3 of the arm, and the measurement will be carried out by the researcher.
Systolic and Diastolic Blood Pressure after the drain removal | 15 minutes after the drain is removed
  After the drain removal blood pressure (mm/Hg) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. Blood Pressure Measurement was performed using a conventional cuffed sphygmomanometer that can measure systolic and diastolic blood pressure, whose reliability was approved according to international standards and calibrated by the company in technical laboratories for certain periods. The cuff of the sphygmomanometer will be inflated to 20 mm / Hg above the systolic pressure by tying it to cover 2/3 of the arm, and the measurement will be carried out by the researcher.
Pulse rate before the drain removal | 15 minutes before the drain removal
  Before the drain removal pulse rate (min) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. The pulse was obtained by the investigator palpating the superficial arteries (by touching them with the hand) and counting the beats felt for one minute. 60 to 100 beats per minute was considered normal for an adult.
Pulse rate as soon as the drain removal | as soon as the drain removal
  As soon as the drain removal pulse rate (min) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. The pulse was obtained by the investigator palpating the superficial arteries (by touching them with the hand) and counting the beats felt for one minute. 60 to 100 beats per minute was considered normal for an adult.
Pulse rate after the drain removal | 15 minutes after the drain is removed
  After the drain removal pulse rate (min) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. The pulse was obtained by the investigator palpating the superficial arteries (by touching them with the hand) and counting the beats felt for one minute. 60 to 100 beats per minute was considered normal for an adult.
Respiration rate before the drain removal | 15 minutes before the drain removal
  Before the drain removal respiration rate (min) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. Respiration rate was measured by the number of diaphragm movements per minute. For an adult at rest, 12 to 20 per minute was considered normal for respiratory rate.
Respiration rate as soon as the drain removal | as soon as the drain removal
  As soon as the drain removal respiration rate (min) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. Respiration rate was measured by the number of diaphragm movements per minute. For an adult at rest, 12 to 20 per minute was considered normal for respiratory rate.
Respiration rate after the drain removal | 15 minutes after the drain is removed
  After the drain removal respiration rate (min) of all patients (lavender oil, cold application, oxygen administration and control group) were measured. Respiration rate was measured by the number of diaphragm movements per minute. For an adult at rest, 12 to 20 per minute was considered normal for respiratory rate.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Urkan, Assoc.Prof., Principal Investigator — Mugla Sıtkı Koçman University
Locations (1):
- Mugla Sitki Kocman University, Muğla, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arıoğlu, B. (2012). The effect of progressive muscle relaxation exercise on pain before chest tube removal. Master's thesis, Çukurova University, Adana.
- [Background] Demir Y, Khorshid L. The effect of cold application in combination with standard analgesic administration on pain and anxiety during chest tube removal: a single-blinded, randomized, double-controlled study. Pain Manag Nurs. 2010 Sep;11(3):186-96. doi: 10.1016/j.pmn.2009.09.002. Epub 2010 May 31. PMID 20728068
- [Background] Tucci G, Amorese V, Romanini E. Closed suction drainage after orthopedic surgery: evidence versus practice. J Orthop Traumatol. 2006; 7: 29-32.
- [Background] Joshi VS, Chauhan S, Kiran U, Bisoi AK, Kapoor PM. Comparison of analgesic efficacy of fentanyl and sufentanil for chest tube removal after cardiac surgery. Ann Card Anaesth. 2007 Jan;10(1):42-5. doi: 10.4103/0971-9784.37923. PMID 17455407
- [Background] Hood BS, Henderson W, Pasero C. Chest tube removal: an expanded role for the bedside nurse. J Perianesth Nurs. 2014 Feb;29(1):53-9. doi: 10.1016/j.jopan.2013.11.001. No abstract available. PMID 24461283
- [Background] Tercan, B. (2015). Nurses' knowledge and application of non-drug methods in pain management. Master's thesis, İnönü University, Malatya.
- [Background] Hsieh LY, Chen YR, Lu MC. Efficacy of cold application on pain during chest tube removal: a randomized controlled trial: A CONSORT-compliant article. Medicine (Baltimore). 2017 Nov;96(46):e8642. doi: 10.1097/MD.0000000000008642. PMID 29145288
- [Background] Ertug N, Ulker S. The effect of cold application on pain due to chest tube removal. J Clin Nurs. 2012 Mar;21(5-6):784-90. doi: 10.1111/j.1365-2702.2011.03955.x. Epub 2011 Nov 15. PMID 22082021
- [Background] Özveren, H. (2011). Non-pharmacological methods in pain control. Faculty of Health Sciences Journal of Nursing, 18 (1), 83-92.
- [Background] Gorji HM, Nesami BM, Ayyasi M, Ghafari R, Yazdani J. Comparison of Ice Packs Application and Relaxation Therapy in Pain Reduction during Chest Tube Removal Following Cardiac Surgery. N Am J Med Sci. 2014 Jan;6(1):19-24. doi: 10.4103/1947-2714.125857. PMID 24678472
- [Background] Gül, A., Eti Aslan, F. (2010). Evidence-Based Approach to Pain Control; Massage and Aromatherapy. Turkey Clinical J Nurs Sci 2012; 4 (1): 30-6
- [Background] Yip YB, Tam AC. An experimental study on the effectiveness of massage with aromatic ginger and orange essential oil for moderate-to-severe knee pain among the elderly in Hong Kong. Complement Ther Med. 2008 Jun;16(3):131-8. doi: 10.1016/j.ctim.2007.12.003. Epub 2008 Mar 4. PMID 18534325
- [Background] Maddocks-Jennings W, Wilkinson JM. Aromatherapy practice in nursing: literature review. J Adv Nurs. 2004 Oct;48(1):93-103. doi: 10.1111/j.1365-2648.2004.03172.x. PMID 15347415
- [Background] Steflitsch W, Steflitsch M. Clinical aromatherapy. Journal of Men's Health 2008; 5 (1): 74-85.
- [Background] Dunning T, James K. Complementary therapies in action--education and outcomes. Complement Ther Nurs Midwifery. 2001 Nov;7(4):188-95. doi: 10.1054/ctnm.2001.0575. PMID 11855801
- [Background] Cooke B, Ernst E. Aromatherapy: a systematic review. Br J Gen Pract. 2000 Jun;50(455):493-6. PMID 10962794
- [Background] Moss M, Cook J, Wesnes K, Duckett P. Aromas of rosemary and lavender essential oils differentially affect cognition and mood in healthy adults. Int J Neurosci. 2003 Jan;113(1):15-38. doi: 10.1080/00207450390161903. PMID 12690999
- [Background] Barocelli E, Calcina F, Chiavarini M, Impicciatore M, Bruni R, Bianchi A, Ballabeni V. Antinociceptive and gastroprotective effects of inhaled and orally administered Lavandula hybrida Reverchon "Grosso" essential oil. Life Sci. 2004 Nov 26;76(2):213-23. doi: 10.1016/j.lfs.2004.08.008. PMID 15519366
- [Background] Kim JT, Wajda M, Cuff G, Serota D, Schlame M, Axelrod DM, Guth AA, Bekker AY. Evaluation of aromatherapy in treating postoperative pain: pilot study. Pain Pract. 2006 Dec;6(4):273-7. doi: 10.1111/j.1533-2500.2006.00095.x. PMID 17129308
- [Background] Braden R, Reichow S, Halm MA. The use of the essential oil lavandin to reduce preoperative anxiety in surgical patients. J Perianesth Nurs. 2009 Dec;24(6):348-55. doi: 10.1016/j.jopan.2009.10.002. PMID 19962101
- [Background] Tulunay, M., Tulunay, F.C. (2000). Pain Assessment and Pain Measurements. Serdar Erdine. (Ed.). In pain (pp. 91-107). Istanbul: Nobel Medical Bookstores.
- [Background] Yazici Sayin Y, Akyolcu N. Comparison of pain scale preferences and pain intensity according to pain scales among Turkish Patients: a descriptive study. Pain Manag Nurs. 2014 Mar;15(1):156-64. doi: 10.1016/j.pmn.2012.08.005. Epub 2012 Sep 24. PMID 24602433
- [Background] Hasanzadeh F, Kashouk NM, Amini S, Asili J, Emami SA, Vashani HB, Sahebkar A. The effect of cold application and lavender oil inhalation in cardiac surgery patients undergoing chest tube removal. EXCLI J. 2016 Jan 22;15:64-74. doi: 10.17179/excli2015-748. eCollection 2016. PMID 27047319
- [Background] Kazan, E.E. (2011). Cold practices and nursing care. Hacettepe University Nursing Faculty Journal, 18 (1), 73-82.
- [Background] Yagiz On A. [Cold applications for the treatment of pain]. Agri. 2006 Apr;18(2):5-14. Turkish. PMID 17089230
- [Background] Love, H.N., Pritchard, K.A., Hart, J.M. ve Saliba, S.A. (2013). Cryotherapy effects, part 1: comparison of skin temperatures and patient-reported sensations for different modes of administration . International Journal of Athletic Therapy and Training, 18(5), 22-30.
- [Background] Steen M, Cooper K, Marchant P, Griffiths-Jones M, Walker J. A randomised controlled trial to compare the effectiveness of ice-packs and Epifoam with cooling maternity gel pads at alleviating postnatal perineal trauma. Midwifery. 2000 Mar;16(1):48-55. doi: 10.1054/midw.1999.0188. PMID 11139861